CLINICAL TRIAL: NCT04488900
Title: A Phase 1, First-in-Human, Double-blind, Randomized, Placebo Controlled Study to Assess the Safety, Tolerability, PK and PD and Food Effect of CKD-508 After Single and Multiple Ascending Oral Dose Administration in Healthy Adult Subjects
Brief Title: Evaluation of the Safety and Tolerability of CKD-508 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A104-01DL2001
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part 1. CKD-508 Capsule in Single Dose (Experimental): Single dose of CKD-508 capsules
  Interventions: Drug: CKD-508 Capsule
- Part 1. Placebo Capsule in Single Dose (Placebo Comparator): Single dose of Placebo capsules
  Interventions: Drug: Placebo Capsule
- Part 2. CKD-508 Tablet in Single Dose (Experimental): Single dose of CKD-508 tablets for biocompartibility
  Interventions: Drug: CKD-508 Tablet
- Part 2. Placebo Tablet in Single Dose (Placebo Comparator): Single dose of Placebo tablets for biocompartibility
  Interventions: Drug: Placebo Tablet
- Part 3. CKD-508 Tablet in Single Dose (Experimental): Single dose of CKD-508 tablets for food effect
  Interventions: Drug: CKD-508 Tablet
- Part 3. Placebo Tablet in Single Dose (Placebo Comparator): Single dose of Placebo tablets for food effect
  Interventions: Drug: Placebo Tablet
- Part 4. CKD-508 Tablet in Multiple Dose (Experimental): Multiple dose of CKD-508 tablets
  Interventions: Drug: CKD-508 Tablet
- Part 4. Placebo Tablet in Multiple Dose (Placebo Comparator): Multiple dose of placebo tablets
  Interventions: Drug: Placebo Tablet

INTERVENTIONS:
Drug: CKD-508 Capsule — Investigational drug
  Arms: Part 1. CKD-508 Capsule in Single Dose
Drug: Placebo Capsule — Placebo
  Arms: Part 1. Placebo Capsule in Single Dose
Drug: CKD-508 Tablet — Investigational drug
  Arms: Part 2. CKD-508 Tablet in Single Dose; Part 3. CKD-508 Tablet in Single Dose; Part 4. CKD-508 Tablet in Multiple Dose
Drug: Placebo Tablet — Placebo
  Arms: Part 2. Placebo Tablet in Single Dose; Part 3. Placebo Tablet in Single Dose; Part 4. Placebo Tablet in Multiple Dose

SUMMARY:
This study is a first-in-human, randomized, placebo-controlled, 4-part, single ascending dose and multiple ascending dose study. The study is designed to assess the safety, tolerability, PK, and PD and food effect of orally administered CKD-508 capsules and tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject voluntarily agrees to participate in this study and signs an Independent Ethics Committee (IEC)-approved informed consent prior to performing any of the Screening Visit procedures.
* Males and females between 18 to 55 years of age, inclusive, at the Screening Visit.
* Females of non-childbearing potential (surgically sterile [hysterectomy or oophorectomy] or postmenopausal (amenorrhea for more than 12 months with follicle-stimulating hormone (FSH) in postmenopausal range confirmed by an FSH test).
* Males must be unable to procreate (defined as surgically sterile [i.e., had a vasectomy ≥6 months prior to screening]) or must agree to use highly effective form of birth control from screening through 90 days after study completion.
* Non-smokers (or other nicotine use) as determined by history (no nicotine use over the past 6 months).

Exclusion Criteria:

* Subject has clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological or psychiatric disorder(s) as determined by the PI or designee.
* Subject has any disorder that would interfere with the absorption, distribution, metabolism or excretion of drugs.
* Subject has any concurrent disease or condition that, in the opinion of the PI, would make the subject unsuitable for participation in the clinical study.
* Subject has history of alcohol and/or illicit drug abuse within 2 years of Screening Visit.
* Subject has positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody or human immunodeficiency virus (HIV) antibody.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2023-07-02 (Actual); Study Completion 2023-07-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability including treatment-emergent AE and treatment-emergent SAE | 28 days post the final dose

SECONDARY OUTCOMES:
Maximum plasma CKD-508 concentrations after dosing | 28 days post the final dose
  Peak plasma concentration (Cmax)
Time of maximum plasma CKD-508 concentrations after dosing | 28 days post the final dose
  Time of peak plasma concentration (Tmax)
Changes from baseline in plasma CKD-508 concentrations in time after dosing | 28 days post the final dose
  Area under the plasma concentration versus time curve (AUC)
Changes from baseline in CETP activity after dosing | 28 days post the final dose
  Pharmacodynamics endpoint
Changes from baseline in lipid parameters after dosing | 14 days post the final dose
  including, but not limited to the following: LDL-C, etc.
  Pharmacodynamics endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Northwick Park Hospital, Harrow, Middlesex, United Kingdom